CLINICAL TRIAL: NCT04381221
Title: Observational Prospective Clinical Feasibility Study of the MyPal ePRO-based Early Palliative Care Digital System in Paediatric Oncology Patients
Brief Title: Observational MyPal-Child Study on the ePRO-based Early Palliative Care Digital System in Paediatric Oncology Patients
Acronym: MyPal4Kids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre for Research and Technology Hellas (Other)
Collaborators: Universität des Saarlandes (Other); Brno University Hospital (Other); Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: MyPal4Kids; DRKS00021458 (Registry Identifier: German Clinical Trials Register); 825872 (Other Grant/Funding Number: Horizon 2020 Grant Agreement Number); U1111-1251-0043 (Registry Identifier: Universal Trial Number (WHO))
Record Dates: First submitted 2020-04-27; First posted 2020-05-08 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Leukemia, Childhood; Solid Tumor, Childhood
Keywords: Patient-Reported Outcome (PRO); electronic Patient-Reported Outcome (ePRO); Patient-Reported Outcome Measure (PROM); Palliative Care for Children; Supportive Care for Children; Serious Game; eHealth; Mobile Applications; Observative Study
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of the study is the evaluation of the feasibility of comprehensive service which has been developed while considering patient-orientated needs. With regard to the study, apps have been developed for both groups of participants, parents and their child which suffers from cancer. These apps aim at supporting the documentation and communication of the own condition. This includes for example a video game which can be played via tablet or smartphone in which questions appear addressing the personally perceived burden by children amongst other things. Participants of the study are children between 6 and 17 years of age which suffer from leukemia or tumors. Further participants of the study are at least one of the patient's parents. It is an observational study. Within the course of the study, the usual treatment is not altered actively by the study, it is, however, supplemented by questionnaires which will be analyzed being anonymized after the end of the study running time.

DETAILED DESCRIPTION:
The study is designed as observational prospective feasibility study. The main objective is to assess the feasibility of a comprehensive, patient-centred service for palliative care in children with cancer by adapting and advancing ePRO systems, which aim at supporting the communication between the patients, their parents and the treating medical healthcare professionals. Participants of the study are pediatric oncology patients between 6 and 17 years of age and at least one of their parents, receiving treatment at one of the participating clinical centers due to leukemia or solid tumors. With regard to the study, apps have been developed for both groups of participants, which includes inter alia a game in which questions about burden considering symptoms can be answered by the children.

ELIGIBILITY:
Inclusion Criteria for Children:

* 6-17 years of age
* Diagnosed with paediatric leukaemia or solid cancer in the past 12 months
* Receiving anti-cancer treatment at one of the participating clinical site
* Have age-appropriate speaking, reading and comprehension skills in either the German or the Czech language
* Provide signed + informed consent from parents or legal representative and the assent form by all children from the age of 14 years. These documents had been evaluated positively by IEC.
* Access to an internet connection and mobile device (e.g. smartphone or tablet)

Inclusion Criteria for Parents:

* Parent(s) with a child eligible for the study, as per the inclusion and exclusion-criteria
* Ability to speak, read and understand German or Czech language
* Provide signed informed consent by parent(s). These documents had been evaluated positively by IEC.
* Access to an internet connection and mobile device (e.g. smartphone or tablet)

Exclusion Criteria for Children:

• Anyone who is not able to participate in the study according to the clinical judgment of the site chief investigator or any other authorized person of the research team. This judgment has to be documented for each child not being enrolled.

Exclusion Criteria for Parents:

• Anyone who is not able to participate in the study according to the clinical judgment of the site chief investigator or any other authorized person of the research team. This judgment has to be documented for each parent not being enrolled.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited in each of the three participating clinical centers. Besides the children patients, an additional group of participants is constituted by the corresponding child's parents. At least one of the parents will be asked to participate in the study as well.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate, defined as percentage of patients eligible for the study from all patients who were screened for the study. | Regularly each month in the course of 6-month course of study enrollment.
  This contributes to the primary study objective: to assess the feasibility and acceptability of a comprehensive, patient-centred service for palliative care and pediatric oncology by adapting and advancing ePRO systems. Further to identify differences between the participating clinical medical centers. This outcome measure also contributes to the secondary objective which is to determine the usage and evaluation of the MyPal apps including the gamified ePRO by children with cancer.
Participation rate, defined as percentage of recruited patients who completed at least 70% of the scheduled questionnaires for 6 months out of all patients eligible for the study | Regularly each month in the course of 6-month course of study enrollment
  This contributes to the primary study objective: to assess the feasibility and acceptability of a comprehensive, patient-centred service for palliative care in children with cancer by adapting and advancing ePRO systems. Further to identify differences between the participating clinical medical centers. This outcome measure also contributes to the secondary objective which is to determine the usage and evaluation of the MyPal apps including the gamified ePRO by children with cancer.
Adherence rate to the different components of the MyPal services by documentation of user behavior and qualitative analysis | Regularly each month in the course of 6-month course of study enrollment
  This contributes to the primary study objective: to assess the feasibility and acceptability of a comprehensive, patient-centred service for palliative care in children with cancer by adapting and advancing ePRO systems. Further to identify differences between the participating clinical medical centers. This outcome measure also contributes to the secondary objective which is to determine the usage and evaluation of the MyPal apps including the gamified ePRO by children with cancer.
Premature discontinuation rate, defined as percentage of recruited patients who have not been followed-up until the end of 6-month course of study enrollment (withdrawal, death or less than 70% completed questionnaires) | Regularly each month in the course of 6-month course of study enrollment
  This contributes to the primary study objective: to assess the feasibility and acceptability of a comprehensive, patient-centred service for palliative care in children with cancer by adapting and advancing ePRO systems. Further to identify differences between the participating clinical medical centers. This outcome measure also contributes to the secondary objective which is to determine the usage and evaluation of the MyPal apps including the gamified ePRO by children with cancer.
System Usability Scale | At the end of the 6-month course of study enrollment
  Min Value: 0, Max Value: 100, higher scores indicate a better outcome. Quantitative data to assess the feasibility and acceptability of a comprehensive, patient-centred service for palliative care in children with cancer by adapting and advancing ePRO systems. Further to identify differences between the participating clinical medical centers. This outcome measure also contributes to the secondary objective which is to determine the usage and evaluation of the MyPal apps including the gamified ePRO by children with cancer.
Structured Interviews and Focus Groups | At the end of the 6-month course of study enrollment
  Qualitative data to assess the feasibility and acceptability of a comprehensive, patient-centred service for palliative care in children with cancer by adapting and advancing ePRO systems. Further to identify differences between the participating clinical medical centers. This outcome measure also contributes to the secondary objective which is to determine the usage and evaluation of the MyPal apps including the gamified ePRO by children with cancer.

SECONDARY OUTCOMES:
Digital adaption of the Mini-SSpedi / SSPedi questionnaires as ePRO. | Once at baseline and several times a week during the 6-month course of study enrollment. The frequency of single questions depends on severity of reported symptom burden.
  Min Value: 0, Max Value: 5, higher scores indicate a worse outcome. To assess children's symptom burden through an in-game ePRO and optionally as standalone ePRO which can be completed outside the serious game.Further, this contributes to the evidence-base of the effectiveness of ePROs in palliative and supportive care for children with cancer.
PedsQL(TM) Cancer Module questionnaire as ePRO. | Once at baseline and each month during the 6-month course of study enrollment.
  Min Value: 0, Max Value: 100, higher scores indicate a better outcome. To demonstrate the appropriateness and acceptability of measures of quality of life of children with cancer.
EORTC PATSAT C-33 questionnaire, adapted appropriately as ePRO to consider parents' perception. | Once at baseline and each month during the 6-month course of study enrollment.
  Min Value: 0, Max Value: 100, higher scores indicate a better outcome. To demonstrate the appropriateness and acceptability of measures of parents' satisfaction with cancer care, i.e. the parents' perception of the quality of medical and nursing care as well as the evaluation of the care's organization and the oncology department services. Furthermore to determine usage and evaluation of the MyPal apps including the gamified ePRO for children with cancer.
Impact on Family Scale questionnaire as ePRO. | Once at baseline and each month during the 6-month course of study enrollment.
  Higher scale scores indicate a worse outcome. To demonstrate the appropriateness and acceptability of measures of the impact of pediatric illness on the family, specifically with regards to financial impact, family-social impact and personal strain.
EQ-5D-3L questionnaire as ePRO. | Once at baseline and each month during the 6-month course of study enrollment.
  Min Value: 11111, Max Value: 33333, higher scores indicate a worse outcome. To demonstrate the appropriateness and acceptability of measures of parents' quality of life having children with cancer. It will be evaluated with regard to the five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Uniquely developed web-based online questionnaire. | Once at the end of the overall course of the study or earlier given the case of changing study staff.
  Higher scores indicate a worse outcome. To determine the impact on health care professionals across Europe due to the integration of ePROs in palliative care by measuring strain parameters etc. caused by the usage of the service which is subject of the study. Furthermore, to contribute to the evidence-base of the effectiveness of ePROs for palliative care for children with cancer

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Stamatopoulos, MD, Study Chair — Representative of the Sponsor: Centre for Research & Technology Hellas; Annette Sander, MD, Principal Investigator — Medical School Hannover; Petr Lokaj, MD, Principal Investigator — University Hospital Brno; Norbert Graf, Professor MD, Study Director — Universität des Saarlandes; Norbert Grad, Professor MD, Principal Investigator — Universität des Saarlandes
Locations (3):
- University Hospital Brno, Brno, Mähren, Czechia
- Germany (2):
  - Medical School Hannover, Hanover, Lower Saxony
  - Saarland University, Homburg, Saarland

IPD SHARING:
Plan to Share IPD: No
The research data will not be published as no consent has been obtained for this. In addition, it is sensitive data derived from a vulnerable patient group, i.e. children in palliative care.
  The research results will only be published in anonymized form and after statistical and qualitative evaluation.
  The study protocol will be published in a scientific journal. The analyses will be conducted until the end of the project. Publications will be made in accordance with the established criteria for publication of the research results, which can be found in the study protocol, as well as in accordance with national data protection guidelines and internationally applicable provisions of the basic data protection regulation.

REFERENCES:
- [Derived] Payne S, Begovic D, Salifu Y, Nelson A, Payne C, Downing J, Natsiavas P, Ling J. Applying Digital Health in Cancer and Palliative Care in Europe: Policy Recommendations from an International Expert Workshop (MyPal Project). J Palliat Med. 2024 Feb;27(2):216-223. doi: 10.1089/jpm.2023.0309. Epub 2023 Sep 22. PMID 37738323
- [Derived] Meyerheim M, Karamanidou C, Payne S, Garani-Papadatos T, Sander A, Downing J, Stamatopoulos K, Ling J, Payne C, Scarfo L, Lokaj P, Maramis C, Graf N. MyPal-Child study protocol: an observational prospective clinical feasibility study of the MyPal ePRO-based early palliative care digital system in paediatric oncology patients. BMJ Open. 2021 Apr 13;11(4):e045226. doi: 10.1136/bmjopen-2020-045226. PMID 33849855
- See also: MyPal project website — https://mypal-project.eu